CLINICAL TRIAL: NCT05932927
Title: Analysis of Clinical Features of Chronic Liver Disease Complicated With Hepatopulmonary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Jie (Other)
Responsible Party: Sponsor-Investigator, Sun Jie, Professor, Beijing YouAn Hospital
Organization: Beijing YouAn Hospital (Other)
Other Study IDs: 2022-096
Record Dates: First submitted 2023-06-09; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Hepatopulmonary Syndrome (HPS)
MeSH Terms: conditions — Hepatopulmonary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic liver disease with hepatopulmonary syndrome: Liver disease (usually cirrhosis with portal hypertension) ；Positive CE-TTE（Contrast enhanced contrast ultrasound）；Abnormal arterial oxygenation: Alveolar-arterial oxygen gradient (AaO2) ≥ 15 mm Hg (>20 mm Hg if age > 64)
  Interventions: Biological: Proteomic sequencing
- Chronic liver disease without hepatopulmonary syndrome: Liver disease (usually cirrhosis with portal hypertension) ； Negative CE-TTE
  Interventions: Biological: Proteomic sequencing

INTERVENTIONS:
Biological: Proteomic sequencing — Proteomic sequencing, bioinformatics analysis，find abnormal indicators between two groups

SUMMARY:
Hepatopulmonary syndrome (HPS) has unknown pathogenesis, limited treatment and poor prognosis. The onset of HPS is insidious and easy to be ignored. Many liver diseases such as "cirrhosis and related complications" are the core characteristics of Beijing You 'an Hospital, but the clinical characteristics of HPS patients in the center are still unclear. The investigators plan to make the diagnosis of HPS among chronic liver disease patients in the hospital according to the diagnostic criteria of HPS proposed in the Practice Guidelines of the International Society of Liver Transplantation in 2016, collect clinical data of HPS participants, evaluate the severity, analyze and summarize clinical characteristics, and conduct management and follow-up. At the same time, The investigators collect blood samples for proteomics tests. In order to improve the diagnosis and treatment level of HPS.

DETAILED DESCRIPTION:
At present, the mechanism of hepatopulmonary syndrome is not clear. The researchers plan to use the extracted plasma for detection, protein extraction and quality control, and then proteolytic hydrolysis, computer detection, and bioinformatics analysis.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis Agreed to venous blood collection

Exclusion Criteria:

* pneumonia, pulmonary vascular disease, interstitial pulmonary disease, COPD, bronchial asthma, lung cancer and other primary pulmonary diseases, acute upper gastrointestinal bleeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver disease admitted to You 'an Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Proteomic results of participants | April 1,2024
  Qualitative and quantitative analysis of proteome

CONTACTS AND LOCATIONS:
Locations (1):
- No.8, Xitoutiao, Youan Men Wai, Fengtai District, Beijing, China